CLINICAL TRIAL: NCT01436578
Title: Post Marketing Surveillance for General Drug Use to Assess the Safety and Efficacy Profile of NOXAFIL Oral Suspension in Usual Practice
Brief Title: Safety and Efficacy of Posaconazole Oral Suspension in Usual Practice in Korea (P08547)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P08547; MK-5592-091 (Other: Merck protocol number)
Record Dates: First submitted 2011-09-16; First posted 2011-09-19 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Fungal Infections
MeSH Terms: conditions — Mycoses | interventions — posaconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: All participants treated with posaconazole oral suspension during the pre-specified surveillance period.
  Interventions: Drug: Posaconazole oral suspension 40 mg/mL

INTERVENTIONS:
Drug: Posaconazole oral suspension 40 mg/mL — Posaconazole oral suspension prescribed according to the current local label
  Other Names: NOXAFIL

SUMMARY:
This study will examine the safety and efficacy of posaconazole in general use in Korea.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

ELIGIBILITY:
Inclusion Criteria:

* Treated with posaconazole oral suspension within current local label

Exclusion Criteria:

* Contraindication to posaconazole oral suspension according to current local label

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants enrolled will be all who are treated with posaconazole oral suspension per the current local label by participating investigators during the pre-specified surveillance period.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2012-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Serious Adverse Experiences | During treatment and for 30 days following cessation of treatment
Number of participants with drug-related adverse experiences | During treatment and for 30 days following cessation of treatment
Number of participants with unexpected drug-related adverse experiences | During treatment and for 30 days following cessation of treatment
Number of participants with Non-Serious Adverse Experiences | During treatment and for 30 days following cessation of treatment
Number of Participants with Responses of Improved, Not Improved, and Worsened | After at least 14 days of treatment